### ALMIRALL, S.A.

# CONFIDENTIAL

When used outside Almirall, S.A.

# **Clinical Trial Protocol Title:**

A MULTICENTER, RANDOMIZED, DOUBLE-BLIND, PARALLEL-GROUP, CONTROLLED STUDY, TO ASSESS THE EFFICACY AND SAFETY OF P-3074 CUTANEOUS SPRAY SOLUTION, IN THE TREATMENT OF MALE PATTERN BALDNESS.



The information contained in this document is the property of Almirall S.A

## Rationale for the amendment

SAP has been amended in order to include a more detailed description of the ITT and the CCI.



Clinical Statistics Page 2 of 3



# 3. Section 8 of the SAP (Changes in Planned Analyses)

## Old text:

**Section 8. Canges in planned analyses** Not applicable

### New text:

## Section 8. Canges in planned analyses

For a better understanding of the ITT population definition, the following wording has been modified:

1- Protocol definition (see section 10.1.1):

ITT population: all patients who will have measurements both at baseline and on treatment

2- SAP definition (see section 5.3):

ITT population: all patients who will have measurements both at baseline and on treatment: i.e. patients who have measurements in regards to hair count both at baseline and on treatment.

| CCI | |
|--------------|---|
| <del>-</del> | |
| | , |

Clinical Statistics Page 3 of 3